CLINICAL TRIAL: NCT01546064
Title: Prospective and Randomized Trial on the Usefulness of T-Tube in the Bile Duct Anastomosis in Liver Transplantation Procedure.
Brief Title: Study to Establish Whether the Use of T-Tube in Bile Duct Anastomosis in Liver Transplantation Decreases Morbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Rafael Lopez Andujar, Head of Unit, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESTUDIOKEHR
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Evidence of Liver Transplantation
Keywords: Bile duct anastomosis; Biliary complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bile duct anastomosis with T-tube (Active Comparator)
  Interventions: Device: Choledocho-choledochostomy with T-tube
- Bile duct anastomosis without T-tube (Active Comparator)
  Interventions: Device: Choledocho-choledochostomy without T-tube

INTERVENTIONS:
Device: Choledocho-choledochostomy with T-tube — In the anastomosis between the common bile duct of the graft and the common bile duct of the recipient, a tutorial T-tube is inserted in the bile duct lumen and will be removed from the patient on third month postoperatively.
  Arms: Bile duct anastomosis with T-tube
Device: Choledocho-choledochostomy without T-tube — The termino-terminal anastomosis between common bile duct of the graft and common bile duct of the recipient is performed without any T-tube.
  Arms: Bile duct anastomosis without T-tube

SUMMARY:
The purpose of this study was to compare the incidence and severity of biliary complications due to liver transplantation after choledochocholedochostomy with or without a T-tube. A per-protocol analysis was designed for recipients of orthotopic liver transplantation in a single center, who were randomly assigned to choledochocholedochostomy with or without a T-tube. It is a prospective and randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a deceased full-size liver graft
* Aged > 18 years

Exclusion Criteria:

* Age < 18 years
* Retransplantation
* Primary sclerosing cholangitis
* Fulminant hepatic failure
* Technical need for a hepaticojejunostomy
* Splitted graft
* Reduced-size graft
* More than one organ transplantation
* Living donation
* Finding of a large difference (twice the size) in common bile duct diameters between the graft and the recipient

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
all morbidity related to bile duct | The first year after liver transplantation procedure
  All the complications related to bile duct that appear after transplantation will be recorded in both groups. All patients will be followed up for the first 12 months after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael López-Andújar, Head of Unit, Principal Investigator — La Fe University and Politechnic Hospital
Locations (1):
- La Fe University and Politechnic Hospital, Valencia, Valencia, Spain

REFERENCES:
- [Background] Duailibi DF, Ribeiro MA Jr. Biliary complications following deceased and living donor liver transplantation: a review. Transplant Proc. 2010 Mar;42(2):517-20. doi: 10.1016/j.transproceed.2010.01.017. PMID 20304182
- [Background] Wojcicki M, Milkiewicz P, Silva M. Biliary tract complications after liver transplantation: a review. Dig Surg. 2008;25(4):245-57. doi: 10.1159/000144653. Epub 2008 Jul 15. PMID 18628624
- [Background] Ayoub WS, Esquivel CO, Martin P. Biliary complications following liver transplantation. Dig Dis Sci. 2010 Jun;55(6):1540-6. doi: 10.1007/s10620-010-1217-2. Epub 2010 Apr 22. PMID 20411422
- [Background] Kizilisik TA, al-Sebayel M, Hammad A, al-Traif I, Ramirez CG. Biliary complications after T-tube placement in liver transplant patients. Transplant Proc. 1997 Nov;29(7):2849-50. doi: 10.1016/s0041-1345(97)00704-5. No abstract available. PMID 9365588
- [Background] Rouch DA, Emond JC, Thistlethwaite JR Jr, Mayes JT, Broelsch CE. Choledochocholedochostomy without a T tube or internal stent in transplantation of the liver. Surg Gynecol Obstet. 1990 Mar;170(3):239-44. PMID 2406979
- [Background] Amador A, Charco R, Marti J, Navasa M, Rimola A, Calatayud D, Rodriguez-Laiz G, Ferrer J, Romero J, Ginesta C, Fondevila C, Fuster J, Garcia-Valdecasas JC. Clinical trial on the cost-effectiveness of T-tube use in an established deceased donor liver transplantation program. Clin Transplant. 2007 Jul-Aug;21(4):548-53. doi: 10.1111/j.1399-0012.2007.00688.x. PMID 17645718
- [Background] Scatton O, Meunier B, Cherqui D, Boillot O, Sauvanet A, Boudjema K, Launois B, Fagniez PL, Belghiti J, Wolff P, Houssin D, Soubrane O. Randomized trial of choledochocholedochostomy with or without a T tube in orthotopic liver transplantation. Ann Surg. 2001 Mar;233(3):432-7. doi: 10.1097/00000658-200103000-00019. PMID 11224633
- [Background] Nuno J, Vicente E, Turrion VS, Pereira F, Ardaiz J, Cuervas V, Barcena R, Garcia M, San Roman AL, Candela A, Honrubia A, Moreno A. Biliary tract reconstruction after liver transplantation: with or without T-tube? Transplant Proc. 1997 Feb-Mar;29(1-2):564-5. doi: 10.1016/s0041-1345(96)00268-0. No abstract available. PMID 9123131
- [Background] Vougas V, Rela M, Gane E, Muiesan P, Melendez HV, Williams R, Heaton ND. A prospective randomised trial of bile duct reconstruction at liver transplantation: T tube or no T tube? Transpl Int. 1996;9(4):392-5. doi: 10.1007/BF00335701. PMID 8819276
- [Background] Sotiropoulos GC, Sgourakis G, Radtke A, Molmenti EP, Goumas K, Mylona S, Fouzas I, Karaliotas C, Lang H. Orthotopic liver transplantation: T-tube or not T-tube? Systematic review and meta-analysis of results. Transplantation. 2009 Jun 15;87(11):1672-80. doi: 10.1097/TP.0b013e3181a5cf3f. PMID 19502959
- [Background] Riediger C, Muller MW, Michalski CW, Huser N, Schuster T, Kleeff J, Friess H. T-Tube or no T-tube in the reconstruction of the biliary tract during orthotopic liver transplantation: systematic review and meta-analysis. Liver Transpl. 2010 Jun;16(6):705-17. doi: 10.1002/lt.22070. PMID 20517904
- [Background] Paes-Barbosa FC, Massarollo PC, Bernardo WM, Ferreira FG, Barbosa FK, Raslan M, Szutan LA. Systematic review and meta-analysis of biliary reconstruction techniques in orthotopic deceased donor liver transplantation. J Hepatobiliary Pancreat Sci. 2011 Jul;18(4):525-36. doi: 10.1007/s00534-010-0346-5. PMID 21127915
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Starzl TE, Putnam CW, Hansbrough JF, Porter KA, Reid HA. Biliary complications after liver transplantation: with special reference to the biliary cast syndrome and techniques of secondary duct repair. Surgery. 1977 Feb;81(2):212-21. PMID 319551
- [Background] Calne RY, McMaster P, Portmann B, Wall WJ, Williams R. Observations on preservation, bile drainage and rejection in 64 human orthotopic liver allografts. Ann Surg. 1977 Sep;186(3):282-90. doi: 10.1097/00000658-197709000-00006. PMID 329780
- [Background] Buczkowski AK, Schaeffer DF, Kim PT, Ho SG, Yoshida EM, Steinbrecher UP, Erb SR, Chung SW, Scudamore CH. Spatulated end-to-end bile duct reconstruction in orthotopic liver transplantation. Clin Transplant. 2007 Jan-Feb;21(1):7-12. doi: 10.1111/j.1399-0012.2006.00556.x. PMID 17302585
- [Background] Neuhaus P, Blumhardt G, Bechstein WO, Steffen R, Platz KP, Keck H. Technique and results of biliary reconstruction using side-to-side choledochocholedochostomy in 300 orthotopic liver transplants. Ann Surg. 1994 Apr;219(4):426-34. doi: 10.1097/00000658-199404000-00014. PMID 8161269
- [Background] Rabkin JM, Orloff SL, Reed MH, Wheeler LJ, Corless CL, Benner KG, Flora KD, Rosen HR, Olyaei AJ. Biliary tract complications of side-to-side without T tube versus end-to-end with or without T tube choledochocholedochostomy in liver transplant recipients. Transplantation. 1998 Jan 27;65(2):193-9. doi: 10.1097/00007890-199801270-00008. PMID 9458013
- [Background] Ben-Ari Z, Neville L, Davidson B, Rolles K, Burroughs AK. Infection rates with and without T-tube splintage of common bile duct anastomosis in liver transplantation. Transpl Int. 1998;11(2):123-6. doi: 10.1007/s001470050115. PMID 9561678
- [Background] Randall HB, Wachs ME, Somberg KA, Lake JR, Emond JC, Ascher NL, Roberts JP. The use of the T tube after orthotopic liver transplantation. Transplantation. 1996 Jan 27;61(2):258-61. doi: 10.1097/00007890-199601270-00017. PMID 8600634
- [Background] Rossi G, Lucianetti A, Gridelli B, Colledan M, Caccamo L, Albani AP, Galmarini M, Fassati LR, Galmarini D. Biliary tract complications in 224 orthotopic liver transplantations. Transplant Proc. 1994 Dec;26(6):3626-8. No abstract available. PMID 7998298
- [Background] Sheng R, Sammon JK, Zajko AB, Campbell WL. Bile leak after hepatic transplantation: cholangiographic features, prevalence, and clinical outcome. Radiology. 1994 Aug;192(2):413-6. doi: 10.1148/radiology.192.2.8029406.
- [Background] Grande L, Perez-Castilla A, Matus D, Rodriguez-Montalvo C, Rimola A, Navasa M, Garcia-Valdecasas JC, Visa J. Routine use of the T tube in the biliary reconstruction of liver transplantation: is it worthwhile? Transplant Proc. 1999 Sep;31(6):2396-7. doi: 10.1016/s0041-1345(99)00398-x. No abstract available. PMID 10500637
- [Background] Rolles K, Dawson K, Novell R, Hayter B, Davidson B, Burroughs A. Biliary anastomosis after liver transplantation does not benefit from T tube splintage. Transplantation. 1994 Feb;57(3):402-4. doi: 10.1097/00007890-199402150-00015. PMID 8108875
- [Background] Bacchella T, Figueira ER, Makdissi FF, Rocha-Santos V, Martino RB, Andraus W, Canedo LF, Machado MA, Machado MC. Biliary reconstruction without T-tube in liver transplantation. Transplant Proc. 2004 May;36(4):951-2. doi: 10.1016/j.transproceed.2004.03.103. PMID 15194330
- [Background] Kusano T, Randall HB, Roberts JP, Ascher NL. The use of stents for duct-to-duct anastomoses of biliary reconstruction in orthotopic liver transplantation. Hepatogastroenterology. 2005 May-Jun;52(63):695-9. PMID 15966185
- [Background] Weiss S, Schmidt SC, Ulrich F, Pascher A, Schumacher G, Stockmann M, Puhl G, Guckelberger O, Neumann UP, Pratschke J, Neuhaus P. Biliary reconstruction using a side-to-side choledochocholedochostomy with or without T-tube in deceased donor liver transplantation: a prospective randomized trial. Ann Surg. 2009 Nov;250(5):766-71. doi: 10.1097/SLA.0b013e3181bd920a. PMID 19809299
- [Background] Shuhart MC, Kowdley KV, McVicar JP, Rohrmann CA, McDonald MF, Wadland DW, Emerson SS, Carithers RL Jr, Kimmey MB. Predictors of bile leaks after T-tube removal in orthotopic liver transplant recipients. Liver Transpl Surg. 1998 Jan;4(1):62-70. doi: 10.1002/lt.500040109. PMID 9457969
- [Background] Koivusalo A, Eskelinen M, Wolff H, Talva M, Makisalo H. Development of T-tube tracts in piglets: effect of insertion method and material of T-tubes. Res Exp Med (Berl). 1997;197(1):53-61. doi: 10.1007/s004330050055. PMID 9226763
- [Background] Apalakis A. An experimental evaluation of the types of material used for bile duct drainage tubes. Br J Surg. 1976 Jun;63(6):440-5. doi: 10.1002/bjs.1800630608. PMID 1276671
- [Background] WINSTONE NE, GOLBY MG, LAWSON LJ, WINDSOR CW. BILIARY PERITONITIS: A HAZARD OF POLYVINYL CHLORIDE T-TUBES. Lancet. 1965 Apr 17;1(7390):843-4. doi: 10.1016/s0140-6736(65)91376-0. No abstract available. PMID 14263542
- [Derived] Lopez-Andujar R, Oron EM, Carregnato AF, Suarez FV, Herraiz AM, Rodriguez FS, Carbo JJ, Ibars EP, Sos JE, Suarez AR, Castillo MP, Pallardo JM, De Juan Burgueno M. T-tube or no T-tube in cadaveric orthotopic liver transplantation: the eternal dilemma: results of a prospective and randomized clinical trial. Ann Surg. 2013 Jul;258(1):21-9. doi: 10.1097/SLA.0b013e318286e0a0. PMID 23426348